CLINICAL TRIAL: NCT04162574
Title: Predicting Binge and Purge Episodes From Passive and Active Apple Watch Data Using a Dynamical Systems Approach
Brief Title: Binge-Eating Genetics Initiative (BEGIN) - Dynamical Systems Approach
Acronym: BEGIN
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Recovery Record (Unknown); University of Utah (Other); uBiome (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-0242; R01MH119084 (NIH)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Binge-Eating Disorder; Bulimia Nervosa
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Saliva samples are collected from each participant for future studies on the genetics of eating disorders
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BEGIN Case: Enrolled participants with BN/BED will participate in a 30-day observational study.
  Interventions: Other: Recovery Record

INTERVENTIONS:
Other: Recovery Record — Observational data will be obtained through participants entering data on disordered eating episodes, mood, and food in Recovery Record, an app to assist people in managing their eating disorder during the 30 days of the trial. In addition, participants wear an Apple Watch from which passive data (e.g., heart rate, activity, and geolocation) are collected.

SUMMARY:
The Binge Eating Genetics Initiative (BEGIN) is an observational study where individuals with binge-eating disorder (BED) or bulimia nervosa (BN) complete assessments about eating disorder history, current disordered eating behavior, and mood. Participants also provide active data on binge eating, purging, nutrition, and cognitions using Recovery Record on the Apple Watch. Passive sensor data are collected via native applications over a 30-day period in 1000 individuals with BED or BN. Investigators will combine longitudinal passive (Apple Watch) and active (Recovery Record) data to predict when patients are at high risk of binge eating or purging. Results will enable the deployment of real-time, in-the-moment, personalized signaling of impending binge or purge episodes that will interrupt automatic behaviors and empower patients to exert control over binge eating and purging by engaging in therapeutic alternatives.

DETAILED DESCRIPTION:
The parent study, BEGIN, has full ethical approval. From within Recovery Record, individuals are directed to a link to the BEGIN study. From outside Recovery Record, interested individuals complete a brief screen. If they are potentially eligible, they are directed to Recovery Record. Informed consent for phenotyping is obtained digitally via the Recovery Record app. After consent, interested participants complete a validated eating disorders diagnostic questionnaire based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria adapted from the Structured Clinical Interview for DSM-5 (ED100K). This questionnaire was developed for use in large genetic studies as a means to recruit large samples efficiently with high diagnostic accuracy. Those who screen case positive are offered the opportunity to participate in the full study (with a second informed consent also delivered from within Recovery Record). Eligible participants are mailed a package containing a description of the study, saliva collection kit, stool collection kit, and an Apple Watch. Participants complete the Eating Disorder Examination Questionnaire (EDE-Q), Generalized Anxiety Disorder 7-item scale (GAD-7), and Patient Health Questionnaire-9 (PHQ-9) at enrollment, midpoint, and endpoint. Participants are asked to log mood and food in the Recovery Record app on their Apple Watch for 30 days, the duration of the study. During those 30-days, participants are also asked to submit their saliva and stool samples. Saliva kits are returned directly to Rutgers University Cell and DNA Repository (RUCDR).

The questionnaire, active, and passive data will all be used to characterize patterns of when and where individuals are more/less likely to binge and/or purge in their daily lives. The investigators will identify low-risk and high-risk passive data patterns that will facilitate the prediction of transitions to high risk states signaling impending binge or purge episodes.

ELIGIBILITY:
Inclusion Criteria:

* Resident of US;
* a current BN or BED diagnosis (confirmed via questionnaire in screening instrument);
* age 18-45 years, inclusive;
* reads, speaks English;
* existing iPhone user with iPhone 5 or later;
* provides informed consent;
* ambulatory

Exclusion Criteria:

* Current use of hormone therapy;
* bariatric surgery, including the following: Roux-en-Y, gastric bypass, laparoscopic adjustable gastric banding, sleeve gastrectomy, duodenal switch with biliopancreatic diversion;
* currently pregnant or breastfeeding;
* thoughts of suicide with a plan in the 2 weeks prior to study enrollment;
* hospitalization due to ED in the 2 weeks prior to study enrollment;
* antibiotic use in the past 30 days (renders temporary ineligibility, but can be - eligible to participate again 30 days after the last dose);
* probiotic use in the past 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals between the ages of 18 and 45, who have an iPhone 5 or later, and who are currently experiencing episodes of binge eating can join the study.
Sampling Method: Non-Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Prediction models for the occurrence of disordered eating episodes in individuals with BN/BED using passive sensor data | all reported disordered eating events during the 30 day observation period
  Dynamic systems approach will use passive and active data to illustrate the dynamics that lead up to a binge or purge event. Using passive data up to two hours prior to a binge or purge event as recorded within the Recovery Record app by the participant (but not within an hour of a previous event), changes in heart rate and actigraphy will be modeled as a function of current heart rate and actigraphy. Time leading up to the binge or purge event, type of event (binge or purge), and an interaction with the type of event will be included as moderators of the relationship of heart and steps in predicting their changes. As one approaches a binge or purge, this will capture a reduction in pattern stability as the strength of association between current heart rate and steps and changes in these same variables should become weaker as one approaches the binge or purge event. This analysis will be able to identify how early signs of instability are detectable before binge and purge events.
Models of the dynamics in the 2 hours after a disordered eating event occurs | all reported disordered eating events during the 30 day observation period
  Using dynamical system approaches, changes in heart rate and steps will be modeled as a function of current levels in heart rate and steps. Time since the binge/purge, type of event, and BN/BED diagnosis (along with interactions between them) will be used as moderators of the relationships of heart rate and actigraphy in predicting the changes.
Prediction models with contextual factors of disordered eating episodes | all reported disordered eating events during the 30 day observation period
  Contextual factors such as positive and negative mood, time of day, prior same day binge eating and/or purging, location, and use of coping skills will be used to inform the models from OUTCOME 1 to see how these factors moderate likelihood of disordered eating episodes. Current mood is assessed within Recovery Record. When participants log a meal, or a binge or purge, they are asked "Which feelings are you experiencing?" There are 28 response options. These include, but are not limited to Happy, Anxious, Lonely, Guilt, Angry, Depressed. Participants can select as many as they like. For each feeling they endorse, they can indicate the level to which they are experiencing these feeling on a 5-point Likert scale, ranging from options such as 'A little' to 'Extreme', where higher values indicate greater intensity of the feeling endorsed.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Bulik, Principal Investigator — UNC at Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and scripts will be made available to the general scientific community at the conclusion of the investigation. Specifically, phenotype data will be submitted to the database of Genotypes and Phenotypes (dbGaP) and National Institute of Mental Health Repository & Genetics Resource (NRGR) and genotype data to dbGaP.
Supporting Information: Study Protocol
Time Frame: Assessment phenotype data will be submitted within 6 months after the end of the study. Genotype data will be submitted after the first set of analyses with these data are complete. All data will be available as long as the repositories maintain the datasets (indefinitely).
Access Criteria: The databases are controlled-access meaning that individuals who wish to have access to the data must apply to the respective repository and meet all of their criteria.
URL: https://nda.nih.gov/get/access-data.html

REFERENCES:
- [Background] Butner JE, Deits-Lebehn C, Crenshaw AO, Wiltshire TJ, Perry NS, Kent de Grey RG, Hogan JN, Smith TW, Baucom KJW, Baucom BRW. A multivariate dynamic systems model for psychotherapy with more than one client. J Couns Psychol. 2017 Nov;64(6):616-625. doi: 10.1037/cou0000238. PMID 29154574
- [Background] Beltz AM, Wright AG, Sprague BN, Molenaar PC. Bridging the Nomothetic and Idiographic Approaches to the Analysis of Clinical Data. Assessment. 2016 Aug;23(4):447-458. doi: 10.1177/1073191116648209. PMID 27165092
- [Background] Butner JE, Wiltshire TJ, Munion AK. Modeling Multi-Agent Self-Organization through the Lens of Higher Order Attractor Dynamics. Front Psychol. 2017 Mar 20;8:380. doi: 10.3389/fpsyg.2017.00380. eCollection 2017. PMID 28373853
- [Background] Butner JE, Gagnon KT, Geuss MN, Lessard DA, Story TN. Utilizing topology to generate and test theories of change. Psychol Methods. 2015 Mar;20(1):1-25. doi: 10.1037/a0037802. Epub 2014 Nov 3. PMID 25365535
- [Derived] Carrino EA, Flatt RE, Pawar PS, Sanzari CM, Tregarthen JP, Argue S, Thornton LM, Bulik CM, Watson HJ. Sociodemographic and clinical characteristics of treated and untreated adults with bulimia nervosa or binge-eating disorder recruited for a large-scale research study. J Eat Disord. 2023 Jul 31;11(1):126. doi: 10.1186/s40337-023-00846-4. PMID 37525298
- [Derived] Igudesman D, Abbaspour A, Reed KK, Flatt RE, Becken B, Thornton LM, Bulik CM, Carroll IM. Laxative Abuse Is Associated With a Depleted Gut Microbial Community Structure Among Women and Men With Binge-Eating Disorder or Bulimia Nervosa: The Binge Eating Genetics Initiative. Psychosom Med. 2023 Oct 1;85(8):727-735. doi: 10.1097/PSY.0000000000001226. Epub 2023 Jun 19. PMID 37363967
- [Derived] Carrino E, Flatt R, Pawar P, Sanzari C, Tregarthen J, Argue S, Thornton L, Bulik C, Watson H. Sociodemographic and Clinical Characteristics of Treated and Untreated Adults with Bulimia Nervosa and/or Binge-eating Disorder Recruited for a Large-Scale Research Study. Res Sq [Preprint]. 2023 May 10:rs.3.rs-2899349. doi: 10.21203/rs.3.rs-2899349/v1. PMID 37214840
- [Derived] Kilshaw RE, Adamo C, Butner JE, Deboeck PR, Shi Q, Bulik CM, Flatt RE, Thornton LM, Argue S, Tregarthen J, Baucom BRW. Passive Sensor Data for Characterizing States of Increased Risk for Eating Disorder Behaviors in the Digital Phenotyping Arm of the Binge Eating Genetics Initiative: Protocol for an Observational Study. JMIR Res Protoc. 2022 Jun 2;11(6):e38294. doi: 10.2196/38294. PMID 35653175
- [Derived] Bulik CM, Butner JE, Tregarthen J, Thornton LM, Flatt RE, Smith T, Carroll IM, Baucom BRW, Deboeck PR. The Binge Eating Genetics Initiative (BEGIN): study protocol. BMC Psychiatry. 2020 Jun 16;20(1):307. doi: 10.1186/s12888-020-02698-7. PMID 32546136